CLINICAL TRIAL: NCT06764121
Title: Impact of Haskalife(TM) Canadian Haskap Berry Powder Formulation on Hypertension and Acuity in Women's Health
Brief Title: Impact of Canadian Haskap Berry Powder on Hypertension and Acuity in Women's Health
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS26475 (B2024:057)
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Hypertension; Alertness
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: The trial will be a 2-period randomized, double-blinded, cross-over study that will last for 16 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither the participants nor the investigators will know the allocation sequence or the identity of the powders.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haskap Powder then Control Powder (Experimental): The participants will consume the haskap powder between weeks 0 and 6. A washout period will occur between weeks 7 and 10. After the washout period, the participants will consume the control powder between weeks 11 and 16. None of the participants or investigators will know the identities of the powder or the participants' allocations.
  Interventions: Other: Haskap Berry Powder; Other: Placebo Powder
- Control Powder then Haskap Powder. (Experimental): The participants will consume the control powder between weeks 0 and 6. A washout period will occur between weeks 7 and 10. After the washout period, the participants will consume the haskap powder between weeks 11 and 16. None of the participants or investigators will know the identities of the powder or the participants' allocations.
  Interventions: Other: Haskap Berry Powder; Other: Placebo Powder

INTERVENTIONS:
Other: Haskap Berry Powder — The participants will consume four packets (16g) of haskap berry powder. The powder can be consumed with other food products.
Other: Placebo Powder — The participants will consume four packets (24g) of placebo powder. The powder can be consumed with other food products.

SUMMARY:
Haskap berries are rich in cyanidin-3-O-glucoside (C3G), which has been shown in vitro to enhance endothelial function. Previous clinical studies suggest haskap berry supplementation may improve cognition, mood, blood pressure, and athletic performance, but research is limited. This trial aims to contribute to the growing body of evidence on the effects of haskap berry supplementation.

The trial is a 2-period, randomized, double-blinded, cross-over design lasting 16 weeks. During the first period (weeks 0-6), participants will receive either haskap berry powder or a control powder. A 4-week washout period follows (weeks 7-10), where no powder is consumed. In the second period (weeks 11-16), participants will receive the powder they did not consume in the first period.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent to participate in the trial;
* Biological female who is at least 35 years of age;
* A waist circumference of at least 35 inches;
* Average systolic blood pressure between 120 and 150 mmHg;
* Average diastolic blood pressure between 75 and 100 mmHg

Exclusion Criteria:

* Biological male;
* Gluten allergies, celiac disease, or gluten intolerance;
* Allergic to berries;
* Receiving chemotherapy;
* Use of medications containing pseudoephedrine or other anti-inflammatory drugs, and the use of cyclosporine or tacrolimusin;
* Cardiovascular diseases including stroke, congestive heart failure, myocardial infarction, unstable angina pectoris, coronary artery bypass graft, percutaneous transluminal coronary angioplasty, and transient ischemic attack within six months before screening;
* Inability to consume treatment product;
* Inability to provide written informed consent;
* Any of the following visual impairments: diabetic retinopathy, age-related macular degeneration, glaucoma, or cataract;
* Risk of epileptic seizures;
* Any form of motor impairments;
* Any visual impairments, uncorrected vision problems, eye disorders, or injuries
* Any medical condition, uncontrolled systemic disease, or concurrent illness that would hinder study compliance or jeopardize the participant's safety, based on the investigator's opinion

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-08-06 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure | Weeks 0, 6, 11, and 16
  The participants' mean awake systolic blood pressure will be measured.

SECONDARY OUTCOMES:
Reaction Time | Weeks 0, 6, 11, and 16
  Mean reaction time to a series of visual stimuli.
Memory | Weeks 0, 6, 11, and 16
  Rey Auditory Verbal Learning Test score
Diastolic Blood Pressure | Weeks 0, 6, 11, and 16
  Mean awake diastolic blood pressure over 3 days
Systolic and Diastolic Blood Pressure | Weeks 0, 6, 11, and 16.
  Mean systolic and diastolic blood pressure measured over three days.
Heart Rate | Weeks 0, 6, 11, and 16
  Mean heart rate measured over three days.

OTHER OUTCOMES:
Acceptability | Weeks 6 and 16
  Overall acceptability of the powder via feedback questionnaire
Clinical Chemistry | Weeks 0, 6, 11, and 16
  Blood Urea Nitrogen, cholesterol, triglycerides, high-density lipoprotein, low-density lipoprotein, fasting blood glucose, creatinine, creatine, albumin, alanine transaminase, and aspartate amino transferase
Weight and waist circumference | Weeks 0, 6, 11, and 16
  Weight (kg) and waist circumference ( inches) will be measured.
Nutritional Intake | Three days before (1) week 0, (2) week 6, (3) week 11, and (4) week 16
  Total calories, carbohydrates, fat, and protein
Physical Activity | Weeks 0, 6, 11, and 16
  The time spent doing (1) vigorous activities, (2) moderate activities, (3) walking, and (4) sedentary activities.
Energy and Mood | Weeks 0, 6, 11, and 16
  Visual analog scale to measure energy and mood

CONTACTS AND LOCATIONS:
Overall Officials: Semone Myrie, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Richardson Centre for Food Technology and Research, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No